CLINICAL TRIAL: NCT04181788
Title: A Phase 1b/2 Open-Label Study to Evaluate Pharmacokinetics, Safety, Efficacy, and Pharmacodynamics of PF-06801591 (PD-1 Inhibitor) in Participants With Advanced Malignancies
Brief Title: Sasanlimab (PF-06801591, PD-1 Inhibitor) in Participants With Advanced Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B8011007; 2019-003818-14 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2019-11-29 (Actual); Results first posted 2023-05-08 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Advanced Malignancies; Non-small-cell Lung Cancer
Keywords: Advanced solid tumors; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm A1 (Phase 1b) (Experimental)
  Interventions: Drug: PF-06801591
- Arm B1 (Phase 1b) (Experimental)
  Interventions: Drug: PF-06801591
- Arm A2 (Phase 2) (Experimental)
  Interventions: Drug: PF-06801591
- Arm B2 (Phase 2) (Experimental)
  Interventions: Drug: PF-06801591

INTERVENTIONS:
Drug: PF-06801591 — A monoclonal antibody (mAb) that blocks the interaction between PD-1 and PDL1/ PD-L2.

SUMMARY:
This is a Phase 1b/2 protocol to evaluate pharmacokinetics, safety, efficacy, and pharmacodynamics of PF-06801591, a programmed death-1(PD-1) antagonist monoclonal antibody (mAb) in participants with advanced malignancies.

This study consists of 2 parts:

Phase 1b part (dose escalation and dose expansion) in patients with advanced malignancies in Asia and a global Phase 2 part in non small cell lung cancer (NSCLC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (≥ 20 years in Japan; ≥ 19 years in South Korea)
* Easter Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate bone marrow function, renal and liver functions Phase 1b
* Histological or Cytological diagnosis of advanced solid tumor with clinical evidence of response to anti-PD-1 or PD-L1 agent
* Participant must have received at least 1 prior line of therapy for recurrent or metastatic disease, and must have progressed/relapsed, be refractory, or intolerant to standard therapy approved for the specific tumor type Phase 2
* Participants must have a documented diagnosis of stage III where participants are not candidates for surgical resection or definitive chemoradiation, or stage IV NSCLC
* EGFR mutation, BRAF mutation, and ALK or ROS1 translocation/rearrangement are not permitted
* Participants whose tumor is known to be PD-L1 positive (Tumor Proportion Score [TPS] ≥1%) or unknown are eligible
* Up to 1 line of prior therapy in advanced or metastatic disease settings allowed
* Participant should not have received prior treatment with anti PD-1/PD-L1 drugs
* At least one measurable lesion as defined by RECIST version 1.1

Exclusion Criteria:

* Participants with known symptomatic brain metastases requiring steroids
* Participants with Interstitial Lung Disease history or complication
* Q-T interval corrected for heart rate QTc > 450 msec for male participants or QTc > 470 msec for female participants or QTc > 480 msec in participants with right bundle branch block.
* Hypertension that cannot be controlled by medications (eg, systolic > 150 mmHg and diastolic > 90 mmHg) despite optimal medical therapy.
* Known or suspected hypersensitivity to active ingredient or excipients of the study drug.
* History of Grade ≥3 immune mediated AE (including AST/ ALT elevations that where considered drug related and cytokine release syndrome [CRS]) that was considered related to prior immune modulatory therapy (eg, immune checkpoint inhibitors, co-stimulatory agents, etc.) and required immunosuppressive therapy (For Phase 1b only).
* Vaccination with live attenuated vaccines within 4 weeks prior to randomization is prohibited; however inactivated vaccines are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2026-06-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (47):
- China (4):
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
- National Cancer Center Hospital, Chuo-ku, Tokyo, Japan
- Russia (19):
  - Russian Research Centre for Radiology and Surgical Technologies, Saint Petersburg, Pesochny
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - Klinika UZI 4D, LLC, Pyatigorsk, Stavropol Kray
  - State budgetary institution of healthcare of Yaroslavl region "Clinical oncology hospital", Yaroslavl, Yaroslavl Oblast
  - Evimed Llc, Chelyabinsk
  - Chelyabinsk Regional Clinical Centre of Oncology and Nuclear Medicine, Chelyabinsk
  - Ars Medika Center, LLC, Kaliningrad
  - GBUZ Regional Clinical Hospital of Kaliningrad region, Kaliningrad
  - Enlimed Llc, Kopeysk
  - Orenburg Regional Clinical Oncological Dispensary, Orenburg
  - Russian Scientific Center For Radiology and Surgical Technologies, Pesochny
  - LLC Medical Center "Magnit", Saint Petersburg
  - Llc "Mss", Saint Petersburg
  - North-West Medical Center, Saint Petersburg
  - Road clinical clinic of JSC "RZD", Saint Petersburg
  - NS HI "Road Clinical Hospital of JSC "Russian Railways"", Saint Petersburg
  - Private Healthcare Institution "Clinical Hospital "RZD-Medicine" of St. Petersburg, Saint Petersburg
  - LLC "Diagnostic center "Energo", Saint Petersburg
  - Medical University REAVIZ, Samara
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Severance Hospital, Yonsei Univ. Health System, Seoul
  - Asan Medical Center, Seoul
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
- Ukraine (17):
  - Limited Liability Company "MedX-ray International Group", Pliuty Village, Kyiv Oblast
  - Asklepion Medical Center, Khodosovka, Kyivska Oblast
  - "Medeya Sumy" LLC, Sumy, Sumska Oblast
  - Communal Non-profit Enterprise City Clinical Hospital #4 of Dnipro City Council, Dnipro
  - Llc "Mdc Expert", Dnipro
  - Municipal Non-profit Enterprise "SubCarpathian Clinical Oncological Centre of Ivano-Frankivsk RC", Ivano-Frankivsk
  - Private Enterprise of Private Manufacturing Company "Acinus", Medical and Diagnostic Center, Kirovohrad
  - Medical centre "Verum" Limited Liability Company, Kyiv
  - Vita Сom LLC, Kyiv
  - The State Institution "Romodanov Neurosurgery Institute,, Kyiv
  - Llc Medical Centre, Odesa
  - Municipal Non-profit Enterprise Odesa Regional Clinical Hospital of Odesa Regional Council, Odesa
  - Llc Lidermed, Odesa
  - Municipal Non Profit enterprise of Sumy Regional Council "Sumy Regional Clinical Oncology Center", Sumy
  - Llc Medical Center Diamed, Uzhhorod
  - MNPE Central City Clinical Hospital of Uzhhorod City Council, Uzhhorod
  - Мunicipal non-profit enterprise "Zhytomyr Regional Oncology Dispensary" of Zhytomyr Regional Council, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Penkov K, Bondarenko I, Saenko DV, Kulyaba Y, Guo J, Gong Y, Yamamoto N, Hotko YS, Boyko V, Fadeeva NV, Ursol GM, Ahn HK, Kislov NV, Shen CI, Davis C, Kowalski K, Michelon E, Pavlov D, Hirohashi T, Cho BC. Pharmacokinetics, safety, and efficacy of an alternative dosing regimen of sasanlimab in participants with advanced NSCLC and other malignancies. Ther Adv Med Oncol. 2024 Sep 11;16:17588359241274592. doi: 10.1177/17588359241274592. eCollection 2024. PMID 39281971
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B8011007

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b Escalation 300 mg SC Q4W: PF-06801591 300 mg was given subcutaneously (SC) every 4 weeks (Q4W) (Cycles are 28 days in length). The maximum number of cycles was 9.
- Phase 1b Expansion 300 mg SC Q4W: PF-06801591 300 mg was given SC Q4W (Cycles are 28 days in length). The maximum number of cycles was 20.
- Phase 1b Escalation 600 mg SC Q6W: PF-06801591 600 mg was given SC every 6 weeks (Q6W) (Cycles are 42 days in length). The maximum number of cycles was 9.
- Phase 1b Expansion 600 mg SC Q6W: PF-06801591 600 mg was given SC Q6W (Cycles are 42 days in length). The maximum number of cycles was 8.
- Phase 2 300 mg SC Q4W: PF-06801591 300 mg was given SC Q4W (Cycles are 28 days in length). The maximum number of cycles was 28.
- Phase 2 600 mg SC Q6W: PF-06801591 600 mg was given SC Q6W (Cycles are 42 days in length). The maximum number of cycles was 18.
Period: TREATMENT
Arm/Group | Phase 1b Escalation 300 mg SC Q4W | Phase 1b Expansion 300 mg SC Q4W | Phase 1b Escalation 600 mg SC Q6W | Phase 1b Expansion 600 mg SC Q6W | Phase 2 300 mg SC Q4W | Phase 2 600 mg SC Q6W
Started | 4 | 12 | 6 | 12 | 41 | 80
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 12 | 6 | 12 | 41 | 80
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 8 | 8
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Progressive disease | 3 | 3 | 5 | 7 | 20 | 38
Not completed — Global deterioration of health status | 0 | 2 | 0 | 0 | 2 | 8
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 3 | 5
Not completed — Other unspecified | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Ongoing | 0 | 3 | 0 | 5 | 7 | 15
Period: FOLLOW-UP
Arm/Group | Phase 1b Escalation 300 mg SC Q4W | Phase 1b Expansion 300 mg SC Q4W | Phase 1b Escalation 600 mg SC Q6W | Phase 1b Expansion 600 mg SC Q6W | Phase 2 300 mg SC Q4W | Phase 2 600 mg SC Q6W
Started (All participants who entered treatment phase were either on-going on treatment or discontinued treatment. Those who discontinued treatment either entered the follow-up period or discontinued the study at the end of treatment.) | 3 | 9 | 6 | 7 | 20 | 49
Completed | 3 | 8 | 4 | 2 | 9 | 22
Not Completed | 0 | 1 | 2 | 5 | 11 | 27
Not completed — Death | 0 | 0 | 1 | 2 | 8 | 20
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other unspecified | 0 | 1 | 0 | 0 | 0 | 3
Not completed — Ongoing | 0 | 0 | 1 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b Escalation 300 mg SC Q4W | Phase 1b Expansion 300 mg SC Q4W | Phase 1b Escalation 600 mg SC Q6W | Phase 1b Expansion 600 mg SC Q6W | Phase 2 300 mg SC Q4W | Phase 2 600 mg SC Q6W | Total
Number analyzed (Participants) | 4 | 12 | 6 | 12 | 41 | 80 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (13.29) | 57.3 (15.78) | 62.7 (10.33) | 62.4 (10.02) | 63.9 (11.75) | 62.9 (10.62) | 62.6 (11.33)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 2 | 7 | 4 | 6 | 18 | 48 | 85
  65 - <75 years | 1 | 5 | 1 | 4 | 17 | 21 | 49
  75 - <85 years | 1 | 0 | 1 | 2 | 5 | 10 | 19
  ≥85 years | 0 | 0 | 0 | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 3 | 9 | 14 | 39
  Male | 0 | 6 | 3 | 9 | 32 | 66 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 12 | 6 | 12 | 41 | 80 | 155
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 0 | 0 | 0 | 34 | 62 | 96
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 12 | 6 | 12 | 7 | 18 | 59
  Multiracial | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with first line (1L) and second line (2L) non-small cell lung cancer (NSCLC) (Phase 2).
  For the Phase 1b, any of the following AEs occurring during the DLT observation period (the first cycle of treatment) which were attributable to the investigational product were classified as DLTs: Grade 5 AE not clearly due to the underlying disease or extraneous causes; Hematologic toxicity; Non-Hematologic Toxicity; Delay of ≥ 3 weeks in receiving the next scheduled administration due to persisting treatment-related toxicities.
Time Frame: Phase 1b: at the end of cycle 1 (28 days) for the PF-06801591 300 mg SC Q4W arms, and (42 days) for the PF-06801591 600 mg SC Q6W arms
Population: DLT-evaluable analysis set included all participants who received at least 1 dose of study treatment in the Phase 1b and either experienced DLT during the DLT-evaluation period or completed the DLT-evaluation period without DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Escalation 300 mg SC Q4W | Phase 1b Expansion 300 mg SC Q4W | Phase 1b Escalation 600 mg SC Q6W | Phase 1b Expansion 600 mg SC Q6W
Number analyzed (Participants) | 3 | 11 | 6 | 12
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 2: AUCτ of PF-06801591 at Steady State
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  AUCτ is area under the plasma concentration-time profile from time zero to the next dose (at steady state, starting at Week 12). (τ = X days, where X = 28 days for Q4W regimen and 42 days for Q6W regimen)
Time Frame: Phase 2: Cycle 4 Day 1, 8, 15, 22 and Cycle 5 Day 1 for the PF-06801591 300 mg SC Q4W arm, and Cycle 3 Day 1, 8, 15, 29 and Cycle 4 Day 1 for the PF-06801591 600 mg SC Q6W arm
Population: Phase 2: The PK concentration analysis set was a subset of the safety analysis set and included participants who had at least 1 reportable concentration measurement. Safety analysis set included all enrolled participants who received at least 1 dose of study drug. Here "Number of participants analyzed" signifies participants who had data available for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*hr/mL)
Arm/Group | Phase 2 300 mg SC Q4W | Phase 2 600 mg SC Q6W
Number analyzed (Participants) | 23 | 49
microgram*hour per milliliter (μg*hr/mL) | 20800 (54) | 48090 (47)
Statistical Analysis 1: Comparison: Phase 2 300 mg SC Q4W vs Phase 2 600 mg SC Q6W; Phase 2 600 mg SC Q6W (experimental) vs. Phase 2 300 mg SC Q4W (control); Test type: Other — Ratio of experimental vs control; Ratio of experimental vs control = 231.20, 90% CI 2-sided [190.09 to 281.21]

3. Primary Outcome: Phase 2: Ctrough of PF-06801591 at Steady State, at Week 12
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  Steady state Ctrough is pre-dose concentration following multiple dosing at steady state (Week 12)
Time Frame: Phase 2: Cycle 4 Day 1 for the PF-06801591 300 mg SC Q4W arm, and Cycle 3 Day 1 for the PF-06801591 600 mg SC Q6W arm
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Phase 2 300 mg SC Q4W | Phase 2 600 mg SC Q6W
Number analyzed (Participants) | 24 | 55
microgram per milliliter (μg/mL) | 21.48 (60) | 23.95 (74)
Statistical Analysis 1: Comparison: Phase 2 300 mg SC Q4W vs Phase 2 600 mg SC Q6W; Phase 2 600 mg SC Q6W (experimental) vs. Phase 2 300 mg SC Q4W (control); Test type: Other — Ratio of experimental vs control; Ratio of experimental vs control = 111.48, 90% CI 2-sided [86.31 to 143.99]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: Phase 1b/2: On-treatment period is defined as the time from the first dose of study treatment through minimum (30 days + last dose of study treatment, start day of new anti-cancer drug therapy - 1 day).
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Laboratory results were classified according to the NCI-CTCAE criteria version 5.0. Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care (ADL); Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Number of participants with Grade 1 to Grade 4 laboratory abnormalities were reported.
Time Frame: as for outcome 4
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Pharmacokinetic Parameters: AUCτ After First Dose
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  AUCτ is area under the plasma concentration-time profile from time zero to the next dose (after single dose). (τ = X days, where X = 28 days for Q4W regimen and 42 days for Q6W regimen)
Time Frame: Phase 1b/2: For the PF-06801591 300 mg SC Q4W arms, Cycle 1 Day 1, 8, 15, 22, Cycle 2 Day 1; for the PF-06801591 600 mg SC Q6W arms, Cycle 1 Day 1, 8, 15, 29, Cycle 2 Day 1
Reporting Status: Not Posted, anticipated posting 2025-12

7. Secondary Outcome: Pharmacokinetic Parameters: Ctrough After First Dose
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  Ctrough is pre-dose concentration after single dose (first dose).
Time Frame: Phase 1b/2: Cycle 2 Day 1 for all Arms
Reporting Status: Not Posted, anticipated posting 2025-12

8. Secondary Outcome: Pharmacokinetic Parameters: Ctrough at Steady State
Description: as for outcome 3
Time Frame: Phase 1b/2: For the PF-06801591 300 mg SC Q4W arms, Day 1 of Cycle 4; for the PF-06801591 600 mg SC Q6W arms, Day 1 of Cycle 3
Reporting Status: Not Posted, anticipated posting 2025-12

9. Secondary Outcome: Number of Participants With Treatment-Induced Anti-Drug Antibody (ADA) /Neutralizing Antibodies (NAb)
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  Treatment-induced ADA = Baseline ADA titer was missing or negative and participant had ≥1 post-treatment positive ADA titer (ADA titer greater than or equal to 99 with assay cut-point of 1.09).
  Treatment-induced NAb = Baseline NAb titer was missing or negative or ADA-negative and participant had ≥1 post-treatment positive NAb titer.
Time Frame: Phase 1b/2: Day 1 of Cycle 1, 2, 3, 4, 6, 8, 10 and end of treatment (EOT) for the PF-06801591 300 mg SC Q4W arms; Day 1 of Cycle 1, 2, 3, 4, 5, 7 and EOT for the PF-06801591 600 mg SC Q6W arms
Reporting Status: Not Posted, anticipated posting 2025-12

10. Secondary Outcome: Number of Participants With Objective Response (OR)
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  OR was defined as confirmed best overall response (BOR) of complete response (CR) or partial response (PR) according to RECIST v1.1.
  Complete Response (CR): Complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). All target lesions must be assessed.
  Partial Response (PR): Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed.
Time Frame: Phase 1b/2: Up to 30 months
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Time to Response (TTR)
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  TTR was defined for participants with confirmed objective response (CR or PR) as the time from the 'start date' to the date of first documentation of objective tumor response which is subsequently confirmed.
Time Frame: Phase 1b/2: Up to 30 months
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: Number of Participants With Objective Response (Complete Response + Partial Response) Reported by Baseline Programmed Death-Ligand 1 (PD-L1) Status (High, Low, and Unknown)
Description: This study included Asian participants with advanced solid tumors (Phase 1b) and global participants with 1L and 2L NSCLC (Phase 2).
  OR was defined as confirmed BOR of CR or PR according to RECIST v1.1. CR: Complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis <10 mm). All target lesions must be assessed.
  PR: Greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. All target lesions must be assessed.
  PD-L1 expression was defined as the number of PD-L1 positive cells and/or qualitative assessment of PD-L1 staining on tumor and inflammatory cells in regions of interest that are defined by tumor cell morphology.
Time Frame: Phase 1b/2: Baseline up to 30 months
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Phase 1b/2: On-treatment period (defined as the time from the first dose of study treatment through minimum [30 days + last dose of study treatment, start day of new anti-cancer drug therapy - 1 day] for the treatment-emergent adverse events (TEAEs); Baseline up to 30 months for all-causality mortality.
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Phase 1b Escalation 300 mg SC Q4W | Phase 1b Expansion 300 mg SC Q4W | Phase 1b Escalation 600 mg SC Q6W | Phase 1b Expansion 600 mg SC Q6W | Phase 2 300 mg SC Q4W | Phase 2 600 mg SC Q6W
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/12 | 1/6 | 2/12 | 16/41 | 31/80
Serious Adverse Events (participants affected / at risk) | 1/4 | 2/12 | 0/6 | 0/12 | 16/41 | 13/80
Other Adverse Events (participants affected / at risk) | 4/4 | 11/12 | 6/6 | 12/12 | 40/41 | 58/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Escalation 300 mg SC Q4W (N=4) | Phase 1b Expansion 300 mg SC Q4W (N=12) | Phase 1b Escalation 600 mg SC Q6W (N=6) | Phase 1b Expansion 600 mg SC Q6W (N=12) | Phase 2 300 mg SC Q4W (N=41) | Phase 2 600 mg SC Q6W (N=80)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inappropriate antidiuretic (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 4 | 2
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 2
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b Escalation 300 mg SC Q4W (N=4) | Phase 1b Expansion 300 mg SC Q4W (N=12) | Phase 1b Escalation 600 mg SC Q6W (N=6) | Phase 1b Expansion 600 mg SC Q6W (N=12) | Phase 2 300 mg SC Q4W (N=41) | Phase 2 600 mg SC Q6W (N=80)
Anaemia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 6 | 8 | 10
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 4 | 3
Supraventricular extrasystoles (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 1 | 5
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 9 | 6
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 5 | 3
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 5 | 3
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 4 | 0
Injection site reaction (General disorders) | 1 | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 1 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 2 | 2
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 3 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 4 | 4
Swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 5
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 1 | 2 | 5 | 6
Amylase increased (Investigations) | 0 | 2 | 0 | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 2 | 4 | 3
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 3 | 2 | 2
Blood corticotrophin decreased (Investigations) | 0 | 1 | 0 | 0 | 2 | 0
Blood corticotrophin increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0 | 2 | 0 | 2
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 4 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 2 | 0 | 1 | 2 | 2
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Cortisol decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Free thyroxine index increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 5
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 3 | 0 | 1 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Thyroid hormones decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Total bile acids increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 0 | 8 | 10
Weight increased (Investigations) | 0 | 2 | 0 | 2 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 2 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 8 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 3 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1 | 2 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 0 | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 4 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 3
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2 | 3
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 6 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 9 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 4 | 3
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 2 | 1 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 3 | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT04181788/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT04181788/SAP_001.pdf